CLINICAL TRIAL: NCT05515185
Title: An Open, Single-arm Clinical Study of Autologous T Cells (CAR-T) Targeting B7-H3 Chimeric Antigen Receptor Gene in the Treatment of Patients With Advanced Gastrointestinal Tumors
Brief Title: B7-H3 Targeting CAR-T Cells Therapy for B7-H3 Positive Solid Tumors
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First People's Hospital of Lianyungang (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KT095
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KT095 CAR-T (Experimental): KT095 CAR-T injection Intravenous infusion
  Interventions: Drug: KT095 CAR-T injection

INTERVENTIONS:
Drug: KT095 CAR-T injection — Clearance of lymphocytes
  Other Names: Fludarabine; Cyclophosphamide

SUMMARY:
This is a clinical study to evaluate the safety and efficacy of CAR-T cells in the treatment of patients with advanced solid tumors in China.

DETAILED DESCRIPTION:
This is a single-center, single-arm, open-label study. This study is planned to enroll about 30 subjects with advanced solid tumors. Autologous CAR-T cells were then infused intravenously into subjects, in a dose-escalating 3+3 design.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70 and of both sexes;
2. Advanced solid tumor diagnosed by histology or pathology;
3. Relapse after receiving chemotherapy or targeted drugs or other second-line therapy;
4. B7H3 antigen was positive in tumor tissues by immunohistochemistry, and the antigen expression rate was more than 15%.
5. Patients had at least one evaluable tumor lesion according to RECIST 1.1 criteria that could be accurately measured at baseline;
6. The ECOG score is 0-2, and the expected survival time is more than 12 weeks;
7. Laboratory test results should at least meet the following requirements:

   Left ventricular ejection fraction ≥40%; Creatinine ≤200 umol/L; Absolute neutrophil count (ANC) ≥1.5×109/L; Platelet (PLT) ≥80×109/L; Hemoglobin ≥80g/L; Oxygen saturation of blood 91%; Total bilirubin ≤2×ULN; ALT and AST 2.5 x ULN or less; The criteria for abnormal ALT and AST due to disease (e.g., liver metastases or bile duct obstruction) or Gilbert syndrome can be relaxed to ≤5×ULN.
8. Having venous access for blood collection or single blood collection;
9. The patient voluntarily participated and signed the informed consent in person.

Exclusion Criteria:

1. pregnant or lactating women;
2. Chemotherapy or radiotherapy was used within 3 days before the blood collection period;
3. Patients who have used systemic steroids within 5 days before blood collection period (except those who have recently or currently used inhaled steroids);
4. Use drugs to stimulate bone marrow hematopoietic cell formation within 5 days before the blood collection period;
5. Those who have used any gene or cell therapy products;
6. History of epilepsy or other central nervous system diseases;
7. Active hepatitis B or C virus, defined as: hepatitis B surface antigen HBsAg or hepatitis B core antibody HBcAb positive subjects with peripheral blood HBV DNA titer above the detection limit; HCV antibody positive for hepatitis C and HCV RNA positive in peripheral blood; People infected with HIV and syphilis;
8. Other tumors in the past 5 years;
9. Patients with severe chest and ascites;
10. There was active or uncontrollable infection requiring systemic treatment within 14 days before enrollment;
11. Other antineoplastic treatments (other than pretreatment and chemotherapy) were administered within 2 weeks before study initiation;
12. The investigator assessed that the patient was unable or unwilling to comply with the protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-09 (Estimated); Primary Completion 2024-09-08 (Estimated); Study Completion 2024-09-08 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | Up to 2 years
  DLT
Maximum tolerable dose | Up to 2 years
  MTD

CONTACTS AND LOCATIONS:
Locations (1):
- Lianyungang First People's Hospital, Lianyungang, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No